CLINICAL TRIAL: NCT02394496
Title: A Randomized Trial With Factorial Design Comparing Fulvestrant ± Lapatinib ± Aromatase Inhibitor in Metastatic Breast Cancer Progressing After Aromatase Inhibitor Therapy
Brief Title: Overcoming Endocrine Resistance in Metastatic Breast Cancer
Acronym: OVER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIM8-OVER; 2007-006031-30 (EudraCT Number)
Record Dates: First submitted 2014-12-16; First posted 2015-03-20 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Fulvestrant; Lapatinib; Aromatase Inhibitor; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Lapatinib; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ARM 1 (Experimental): Fulvestrant + Placebo Lapatinib
  Interventions: Drug: Fulvestrant; Drug: Placebo Lapatinib
- ARM 2 (Experimental): Fulvestrant + Aromatase Inhibitors + Placebo Lapatinib
  Interventions: Drug: Fulvestrant; Drug: Aromatase Inhibitors; Drug: Placebo Lapatinib
- ARM 3 (Experimental): Fulvestrant + Lapatinib
  Interventions: Drug: Fulvestrant; Drug: Lapatinib
- ARM 4 (Experimental): Fulvestrant + Lapatinib + Aromatase Inhibitors
  Interventions: Drug: Fulvestrant; Drug: Lapatinib; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500mg (2 x 5ml) im injections as a loading dose on Day 0, followed by 500mg (2x5ml) on Day 14 (+/- 3 days) , Day 28 (+/- 3 days) and every 28 Days (+/- 3 days) thereafter.
  Other Names: Faslodex
Drug: Lapatinib — 1500mg (TBD) O.S. qd
  Arms: ARM 3; ARM 4
Drug: Aromatase Inhibitors — as indicated in the Summary Product Characteristic
  Other Names: Aromatase Inhibitor
  Arms: ARM 2; ARM 4
Drug: Placebo Lapatinib — 1500mg (TBD) O.S. qd
  Other Names: Placebo
  Arms: ARM 1; ARM 2

SUMMARY:
Based on these results it can be envisioned that the majority of endocrine-responsive post-menopausal breast cancer patients will be treated with an AI as adjuvant therapy (front-line, switching or extending) and/or as first-line management of metastatic breast cancer.

DETAILED DESCRIPTION:
In presence of ER hypersensitivity even a small amount of ER may be sufficient for sustained growth signalling. On the other hand, ER disruption operated by fulvestrant is not complete, particularly in the initial phase of treatment. From phase III trials, indeed, The invertigators know that with the standard 250mg monthly dose the steady state of circulating drug is reached only after 5-6 injections. This may play a role since, as long as ER downregulation is concerned, a clear dose-response relationship has been reported. In such a situation, fulvestrant efficacy may be partial, particularly because the concomitant AI discharge yields a restoration of physiologic postmenopausal levels of circulating oestrogens. New dosing schedule are currently under investigation both to accelerate the achievement of the steady state (loading dose) and to achieve higher circulating drug levels (high dose) (86).

In this trial the investigators will be using the so-called 'loading dose'.

Further potential strategies to improve fulvestrant efficacy in this setting are:

A) avoid the restoration of circulating oestrogens; B) interfere with molecular mechanisms that produce ER hypersensitivity by targeting the EGFR/ERBB2/ERB3 system.

A) avoid the restoration of circulating oestrogens: this should be achieved by holding the AI treatment. Because some cases of progression upon AIs may be related to an inefficient inhibition of the aromatase it is a logical step to test whether changing AI class (from type I, steroidal, to type II, non steroidal, and vice-versa) (87), may improve fulvestrant efficay. In this view, pts in this trial will be randomized to receive fulvestrant (loading dose) with or without the alternate class AI treatment. Circulating oestrogens levels will be tracked to verify inhibition of aromatase for pts assigned to concurrent AI treatment.

B) Interfere with growth factors-mediated ER hypersensitivity: although fulvestrant is able to overcome the ER hypersensitivity of LTED (88) and produce a growth arrest, this activity may not be complete because of incomplete ER disruption, but also because of a direct stimulation of growth by the hyperactivated EGFR/ERBB2/ERB3 system. Laboratory evidence support this hypothesis. Indeed, breast cancer cell lines exposed to long-term treatment with fulvestrant became insensitive to the drug and restore growth (89). This growth does not appear, however, related to the development of direct resistance to the drug, since ER mediated signalling continue to be efficiently suppressed in these cells; rather it may be driven by the use of alternative growth-stimulating pathway, including the EGFR system. Indeed, it can be abrogated by the EGFR-tyrosine Kinase inhibitor Gefitinib (IRESSA™) and by an MAPK-inhibitor (90). Lapatinib (GW572016) is an orally active small molecule that reversibly inhibits ErbB1 and ErbB2 tyrosine kinases, which in turn blocks phosphorylation and activation of Erk1/2 (p-Erk1/2) and Akt (p-Akt) in ErbB1- and/ or ErbB2-expressing tumor cell lines and xenografts (91-94). Lapatinib elicits cytostatic or cytotoxic antitumor effects depending on the cell type (95;96). Because ErbB2-containing heterodimers exert potent mitogenic signals, simultaneously interrupting both ErbB1 and ErbB2 signaling is an appealing therapeutic approach. Moreover, ErbB3 signaling is also involved in lapatinib action. Indeed ErbB3 is kinase-dead and relies on ErbB2 for transactivation: ErbB2-ErbB3 heterodimers are potent activators of the PI3K-Akt survival pathway (97;98), which can, in turn, inhibited by lapatinib.

Based on its molecular mechanism of action, on its fair toxicity profile and on its promising, although preliminary, activity data, Lapatinib appears an ideal candidate to combine with Fulvestrant in the attempt to improve its efficacy in patients progressing on AIs.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Histological/cytological confirmation of breast cancer
3. Documented positive hormone receptor status (ER+ve and/or PgR+ve) of primary or metastaic tumor issue, according to the local laboratory parameters
4. Postmenopausal women
5. Confirmed progression of disease after an adjuvant therapy or a therapy for metastatic disease with an aromatase inhibitors
6. Patients demonstrating prior response to AI therapy
7. Patients with measurable disease as per RECIST criteria /Patients with bone lesions, lytic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST criteria.
8. May have received prior radiotherapy as treatment for primary or metastatic tumour; however, is not required for study entry;
9. Life expectancy of at least 8 months
10. WHO performance status 0, 1 or 2
11. Patients with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence.
12. Are able to swallow and retain oral medication;
13. Are able to complete all screening assessments as outlined in the protocol;
14. Patients must have normal organ and marrow function
15. Left ventricular ejection fraction (LVEF) within the institutional normal range

Exclusion Criteria:

1. Previous therapy with Fulvestrant and/or Lapatinib;
2. Patients with HER 2 overexpressing, either IHC 3+ or FISH +;
3. Concurrent non study anti-cancer therapy (
4. Have unresolved or unstable, serious toxicity from prior administration
5. Have malabsorption syndrome,
6. Have a concurrent disease or condition that would make the patient inappropriate for study participation,
7. Have an active or uncontrolled infection;
8. Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
9. Have a known history of uncontrolled or symptomatic angina, arrhythmias, or CHF;
10. Receive concurrent treatment with an investigational agent or participate in another clinical trial;
11. Receive concurrent treatment with prohibited medications
12. Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication;
13. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to fulvestrant, aromatase inhibitors or lapatinib or excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2007-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  Progression free survival (PFS): it is defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time To Progression | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  Time to Progression (TTP): it is defined as the time between the first study dose administration and the date of progression of the disease or cancer-related death, whichever occurs first.
Overall Survival | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  Overall survival. (OS): it is defined as the time between the first study dose administration and the date death from any cause.
Response Rate: | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  Response Rate: It will be classified according to the RECIST criteria.
Clinical Benefit Rate | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 6 months
  Clinical Benefit Rate: it is defined as the sum of rates of PR, CR and SD lasting ≥ 6 months.
Safety as measured by expected and Non-expected toxicity events | Defined as the time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  To evaluate expected and Non-expected toxicity events that occur in more than 5% of patients in any of the study group, as reported by the CTC.
Safety assessed by number of Participants with Adverse Events | time between the first study dose administration and the date of progression of the disease or death from any cause, whichever occurs first assessed up to 12 months
  Withdrawals from the treatment plan (causes of withdrawals will be compared per each study group).

CONTACTS AND LOCATIONS:
Overall Officials: Sabino De Placido, MD, Principal Investigator — Dipartimento di Medicina Clinica e Chirurgia Oncologia Università degli Studi di Napoli "Federico II"; Michelino De Laurentiis, MD, Study Chair — Istituto Nazionale dei Tumori - Fondazione G. Pascale
Locations (69):
- Italy (69):
  - A.S.U.R. Zona Territoriale 6 Fabriano U.O. Oncologia Medica, Fabriano, Ancona
  - Istituto Tumori 'Giovanni Paolo II' - IRCCS Ospedale Oncologico U.O. Oncologia Medica e Sperimentale, Bari, Bari
  - Azienda Ospedaliera G. Rummo U.O. di Oncologia Medica, Benevento, Benevento
  - Ospedale Fatebenefratelli 'Sacro Cuore di Gesù' U.O. Oncologia, Benevento, Benevento
  - Azienda Ospedaliera Treviglio-Caravaggio U.O. Oncologia Medica, Treviglio, Bergamo
  - Presidio Ospedaliero 'Antonio Perrino' U.O.C. di Oncologia, Brindisi, Brindisi
  - dazione di Ricerca e Cura 'Giovanni Paolo II' U.O. di Ginecologia Oncologia, Campobasso, Campobasso
  - Ospedale Civile di Campobasso - A. Cardarelli U.O.C. Oncologia Medica, Campobasso, Campobasso
  - Azienda Ospedaliera 'Sant'Anna e San Sebastiano' U.O.C. di Oncologia, Caserta, Caserta
  - Presidio Ospedaliero Garibaldi - Nesima S.C. di Oncologia Medica, Catania, Catania
  - A.O.U. Ospedale Vittorio Emanuele e Ferrarotto U.O. di Oncologia Medica, Catania, Catania
  - Humanitas Centro Catanese di Oncologia U.O. Oncologia Medica, Catania, Catania
  - Ospedale Civile Renzetti U.O. Oncologia Medica, Lanciano, Chieti
  - Azienda Ospedaliera S. Anna U.O. di Oncologia Medica, Como, Como
  - Ospedale S. Francesco da Paola U.O. Oncologia Medica, Paola, Cosenza
  - Arcispedaliera S. Anna di Ferrara U.O. Oncologia Clinica, Ferrara, Ferrara
  - IRCCS - 'Casa Sollievo della Sofferenza' U.O. Oncologia Medica, San Giovanni Rotondo, Foggia
  - Ospedale 'SS. Trinità' U.O. Oncologia Medica, Sora, Frosinone
  - I.R.C.C.S. A.O.U. San Martino - I.S.T. S.C. Oncologia Medica A, Genova, Genova
  - ASRM - Ospedale F. Veneziale - Zona di Isernia U.O. Oncologia, Isernia, Isernia
  - A.S.L. LT - Ospedale Santa Maria Goretti U.O.C. di Oncologia Medica, Latina, Latina
  - Ospedale Vito Fazzi U.O. di Oncologia, Lecce, Lecce
  - Ospedale Unico Versilia U.O. Oncologia Medica, Lido di Camaiore, Lucca
  - Ospedale Civico San Vincenzo U.O. Oncologia Medica, Taormina, Messina
  - Istituto Europeo di Oncologia (IRCCS) Dipartimento di Medicina - Unità Cure Mediche, Milan, Milano
  - Azienda Ospedaliera Cardarelli Divisione Di Oncologia, Napoli, Napoli
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale U.O. Oncologia Medica Senologica, Napoli, Napoli
  - Università di Napoli Federico II - Facoltà di Medicina Dipartimento di Medicina Clinica e Chirurgia - Oncologia, Napoli, Napoli
  - A.O.U. 'Maggiore della Carità' S.C. Oncologia, Novara, Novara
  - Istituto Oncologico Veneto - I.R.C.C.S. U.O. di Oncologia Medica II, Padua, Padova
  - A.O.U.P. 'Paolo Giaccone' U.O.C. di Oncologia Medica, Palermo, Palermo
  - A.R.N.A.S - Ospedale Civico e Benfratelli G. Di Cristina e M. Ascoli Divisione di Oncologia Medica, Palermo, Palermo
  - Fondazione S. Maugeri IRCCS U.O. Oncologia Medica II, Pavia, Pavia
  - IRCCS Policlinico S. Matteo S.C. di Oncologia Medica, Pavia, Pavia
  - Ospedale S. Maria della Misericordia S.C. Oncologia Medica, Perugia, Perugia
  - AUSL di Piacenza - Ospedale U.O. Oncologia Medica, Piacenza, Piacenza
  - Ospedale 'Felice Lotti' - Azienda USL 5 di Pisa U.O. di Oncologia Medica, Pontedera, Pisa
  - Centro di Riferimento Oncologico S.O.C. di Oncologia Medica C, Aviano, Pordenone
  - Azienda Ospedaliera Santa Maria degli Angeli U.O. Oncolgia Medica, Pordenone, Pordenone
  - Ospedale Oncologico Regionale - Centro di Riferimento Oncologico di Basilicata U.O. di Oncologia Medica, Rionero in Vulture, Potenza
  - Azienda Ospedaliera Bianchi - Melacrino - Morelli U.O. di Oncologia Medica, Reggio Calabria, Reggio Calabria
  - Ospedale San Sebastiano Day Hospital Oncologico - Divisione Medicina Acuti, Correggio, Reggio Emilia
  - Arcispedale S.Maria Nuova Servizio di Oncologia, Reggio Emilia, Reggio Emilia
  - Istituto Regina Elena per lo studio e la cura dei tumori S.C. Oncologia Medica A, Roma, Roma
  - Azienda Ospedaliera San Camillo - Forlanini Day Hospital Oncologia Mammella, Roma, Roma
  - Policlinico Universitario 'Agostino Gemelli' U.O.C. Ginecologia Oncologica, Roma, Roma
  - Ospedale Fatebenefratelli San Giovanni Calibita - Isola Tiberina U.O. Oncologia, Roma, Roma
  - Azienda Ospedaliera S. Andrea - Università La Sapienza U.O.C. Oncologia, Roma, Roma
  - Ospedale San Pietro Fatebenefratelli Dipartimento di Oncologia - Day Hospital Oncologico, Roma, Roma
  - Azienda Ospedaliera - Ospedale Umberto I U.O. di Medicina e Oncoematologia, Nocera Inferiore, Salerno
  - Ospedale G. Da Procida - ASL SA U.O. di Oncologia, Salerno, Salerno
  - Azienda Ospedaliera 'San Giovanni di Dio e Ruggi D'Aragona' Struttura Complessa di Oncologia, Salerno, Salerno
  - Presidio Ospedaliero di Vallo della Lucania U.O. Oncologia Medica, Vallo della Lucania, Salerno
  - Azienda Ospedaliera n. 1 - Annunziata Oncologia Medica, Sassari, Sassari
  - Università di Sassari U.O. di Oncologia Medica, Sassari, Sassari
  - AOVV - Ospedale E. Morelli S.O.C. Medicina Interna - D.H. Oncologico-Ematologico-Internistico, Sondalo, Sondrio
  - Ospedale Civile di Sondrio - Azienda Ospedaliera Valtellina e Valchiavenna S.C. Oncologia Medica, Sondrio, Sondrio
  - Fondazione del Piemonte per l'Oncologia - Istituto di Ricovero e Cura a Carattere Scientifico (I.R.C.C.S.) Direzione di Oncologia Medica, Candiolo, Torino
  - Ospedale Evangelico Valdese - ASL TO1 U.O. di Oncologia Medica, Torino, Torino
  - Presidio San Lazzaro - A.O.U. San Giovanni Battista di Torino (Molinette) S.C. Oncologia Medica II, Torino, Torino
  - Università degli Studi di Torino - Ospedale S. Anna U.O. di Oncologia Medica, Torino, Torino
  - Ospedale Mauriziano Umberto I S.C.D.U. Ginecologia e Ostetricia, Torino, Torino
  - Centro Oncologico A.S.S. N°1 Triestina Centro Sociale Oncologico, Trieste, Trieste
  - A.O.U. ´S. Maria della Misericordia´ Dipartimento di Oncologia, Udine, Udine
  - Ospedale 'S. Antonio Abate' U.O. Oncologia, Gallarate, Varese
  - Azienda Ospedaliera Busto Arsizio - Presidio Ospedaliero Saronno S.C. Oncologia Medica, Saronno, Varese
  - Azienda Ospedaliera Circolo e Fondazione Macchi U.O. di Oncologia Medica, Varese, Varese
  - Ospedale Sacro Cuore - Don Calabria U.O.C. Oncologia Medica, Negrar, Verona
  - Presidio Ospedaliero 'Belcolle' U.O.C. Oncologia Medica, Viterbo, Viterbo

REFERENCES:
- [Background] McPherson K, Steel CM, Dixon JM. ABC of breast diseases. Breast cancer-epidemiology, risk factors, and genetics. BMJ. 2000 Sep 9;321(7261):624-8. doi: 10.1136/bmj.321.7261.624. No abstract available. PMID 10977847
- [Background] Fisher B, Anderson S, Tan-Chiu E, Wolmark N, Wickerham DL, Fisher ER, Dimitrov NV, Atkins JN, Abramson N, Merajver S, Romond EH, Kardinal CG, Shibata HR, Margolese RG, Farrar WB. Tamoxifen and chemotherapy for axillary node-negative, estrogen receptor-negative breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-23. J Clin Oncol. 2001 Feb 15;19(4):931-42. doi: 10.1200/JCO.2001.19.4.931. PMID 11181655
- [Background] Meric F, Hung MC, Hortobagyi GN, Hunt KK. HER2/neu in the management of invasive breast cancer. J Am Coll Surg. 2002 Apr;194(4):488-501. doi: 10.1016/s1072-7515(02)01121-3. No abstract available. PMID 11949754
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Nicholson RI, Gee JM, Harper ME. EGFR and cancer prognosis. Eur J Cancer. 2001 Sep;37 Suppl 4:S9-15. doi: 10.1016/s0959-8049(01)00231-3. PMID 11597399
- [Background] Yarden Y, Sliwkowski MX. Untangling the ErbB signalling network. Nat Rev Mol Cell Biol. 2001 Feb;2(2):127-37. doi: 10.1038/35052073. PMID 11252954
- [Background] Burstein HJ. The distinctive nature of HER2-positive breast cancers. N Engl J Med. 2005 Oct 20;353(16):1652-4. doi: 10.1056/NEJMp058197. No abstract available. PMID 16236735
- [Background] Lu Y, Zi X, Zhao Y, Mascarenhas D, Pollak M. Insulin-like growth factor-I receptor signaling and resistance to trastuzumab (Herceptin). J Natl Cancer Inst. 2001 Dec 19;93(24):1852-7. doi: 10.1093/jnci/93.24.1852. PMID 11752009
- [Background] Xia W, Liu LH, Ho P, Spector NL. Truncated ErbB2 receptor (p95ErbB2) is regulated by heregulin through heterodimer formation with ErbB3 yet remains sensitive to the dual EGFR/ErbB2 kinase inhibitor GW572016. Oncogene. 2004 Jan 22;23(3):646-53. doi: 10.1038/sj.onc.1207166. PMID 14737100
- [Background] Gerber HP, Malik AK, Solar GP, Sherman D, Liang XH, Meng G, Hong K, Marsters JC, Ferrara N. VEGF regulates haematopoietic stem cell survival by an internal autocrine loop mechanism. Nature. 2002 Jun 27;417(6892):954-8. doi: 10.1038/nature00821. PMID 12087404
- [Background] Albanell J, Codony-Servat J, Rojo F, Del Campo JM, Sauleda S, Anido J, Raspall G, Giralt J, Rosello J, Nicholson RI, Mendelsohn J, Baselga J. Activated extracellular signal-regulated kinases: association with epidermal growth factor receptor/transforming growth factor alpha expression in head and neck squamous carcinoma and inhibition by anti-epidermal growth factor receptor treatments. Cancer Res. 2001 Sep 1;61(17):6500-10. PMID 11522647
- [Background] Rubin Grandis J, Melhem MF, Gooding WE, Day R, Holst VA, Wagener MM, Drenning SD, Tweardy DJ. Levels of TGF-alpha and EGFR protein in head and neck squamous cell carcinoma and patient survival. J Natl Cancer Inst. 1998 Jun 3;90(11):824-32. doi: 10.1093/jnci/90.11.824. PMID 9625170
- [Background] Howell GM, Humphrey LE, Awwad RA, Wang D, Koterba A, Periyasamy B, Yang J, Li W, Willson JK, Ziober BL, Coleman K, Carboni J, Lynch M, Brattain MG. Aberrant regulation of transforming growth factor-alpha during the establishment of growth arrest and quiescence of growth factor independent cells. J Biol Chem. 1998 Apr 10;273(15):9214-23. doi: 10.1074/jbc.273.15.9214. PMID 9535913
- [Background] Jiang D, Yang H, Willson JK, Liang J, Humphrey LE, Zborowska E, Wang D, Foster J, Fan R, Brattain MG. Autocrine transforming growth factor alpha provides a growth advantage to malignant cells by facilitating re-entry into the cell cycle from suboptimal growth states. J Biol Chem. 1998 Nov 20;273(47):31471-9. doi: 10.1074/jbc.273.47.31471. PMID 9813060
- [Background] Rusnak DW, Affleck K, Cockerill SG, Stubberfield C, Harris R, Page M, Smith KJ, Guntrip SB, Carter MC, Shaw RJ, Jowett A, Stables J, Topley P, Wood ER, Brignola PS, Kadwell SH, Reep BR, Mullin RJ, Alligood KJ, Keith BR, Crosby RM, Murray DM, Knight WB, Gilmer TM, Lackey K. The characterization of novel, dual ErbB-2/EGFR, tyrosine kinase inhibitors: potential therapy for cancer. Cancer Res. 2001 Oct 1;61(19):7196-203. PMID 11585755
- [Background] Vogel CL, Cobleigh MA, Tripathy D, Gutheil JC, Harris LN, Fehrenbacher L, Slamon DJ, Murphy M, Novotny WF, Burchmore M, Shak S, Stewart SJ, Press M. Efficacy and safety of trastuzumab as a single agent in first-line treatment of HER2-overexpressing metastatic breast cancer. J Clin Oncol. 2002 Feb 1;20(3):719-26. doi: 10.1200/JCO.2002.20.3.719. PMID 11821453
- [Background] Grossi PM, Ochiai H, Archer GE, McLendon RE, Zalutsky MR, Friedman AH, Friedman HS, Bigner DD, Sampson JH. Efficacy of intracerebral microinfusion of trastuzumab in an athymic rat model of intracerebral metastatic breast cancer. Clin Cancer Res. 2003 Nov 15;9(15):5514-20. PMID 14654531
- [Background] Pestalozzi BC, Brignoli S. Trastuzumab in CSF. J Clin Oncol. 2000 Jun;18(11):2349-51. doi: 10.1200/JCO.2000.18.11.2349. No abstract available. PMID 10829059
- [Background] Cobleigh MA, Vogel CL, Tripathy D, Robert NJ, Scholl S, Fehrenbacher L, Wolter JM, Paton V, Shak S, Lieberman G, Slamon DJ. Multinational study of the efficacy and safety of humanized anti-HER2 monoclonal antibody in women who have HER2-overexpressing metastatic breast cancer that has progressed after chemotherapy for metastatic disease. J Clin Oncol. 1999 Sep;17(9):2639-48. doi: 10.1200/JCO.1999.17.9.2639. PMID 10561337
- [Background] Burstein HJ, Kuter I, Campos SM, Gelman RS, Tribou L, Parker LM, Manola J, Younger J, Matulonis U, Bunnell CA, Partridge AH, Richardson PG, Clarke K, Shulman LN, Winer EP. Clinical activity of trastuzumab and vinorelbine in women with HER2-overexpressing metastatic breast cancer. J Clin Oncol. 2001 May 15;19(10):2722-30. doi: 10.1200/JCO.2001.19.10.2722. PMID 11352965
- [Background] Bendell JC, Domchek SM, Burstein HJ, Harris L, Younger J, Kuter I, Bunnell C, Rue M, Gelman R, Winer E. Central nervous system metastases in women who receive trastuzumab-based therapy for metastatic breast carcinoma. Cancer. 2003 Jun 15;97(12):2972-7. doi: 10.1002/cncr.11436. PMID 12784331
- [Background] Clayton AJ, Danson S, Jolly S, Ryder WD, Burt PA, Stewart AL, Wilkinson PM, Welch RS, Magee B, Wilson G, Howell A, Wardley AM. Incidence of cerebral metastases in patients treated with trastuzumab for metastatic breast cancer. Br J Cancer. 2004 Aug 16;91(4):639-43. doi: 10.1038/sj.bjc.6601970. PMID 15266327
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Encarnacion CA, Ciocca DR, McGuire WL, Clark GM, Fuqua SA, Osborne CK. Measurement of steroid hormone receptors in breast cancer patients on tamoxifen. Breast Cancer Res Treat. 1993;26(3):237-46. doi: 10.1007/BF00665801. PMID 8251648
- [Background] Hull DF 3rd, Clark GM, Osborne CK, Chamness GC, Knight WA 3rd, McGuire WL. Multiple estrogen receptor assays in human breast cancer. Cancer Res. 1983 Jan;43(1):413-6. PMID 6847780
- [Background] Buzdar AU, Jonat W, Howell A, Jones SE, Blomqvist CP, Vogel CL, Eiermann W, Wolter JM, Steinberg M, Webster A, Lee D. Anastrozole versus megestrol acetate in the treatment of postmenopausal women with advanced breast carcinoma: results of a survival update based on a combined analysis of data from two mature phase III trials. Arimidex Study Group. Cancer. 1998 Sep 15;83(6):1142-52. PMID 9740079
- [Background] Buzdar A, Douma J, Davidson N, Elledge R, Morgan M, Smith R, Porter L, Nabholtz J, Xiang X, Brady C. Phase III, multicenter, double-blind, randomized study of letrozole, an aromatase inhibitor, for advanced breast cancer versus megestrol acetate. J Clin Oncol. 2001 Jul 15;19(14):3357-66. doi: 10.1200/JCO.2001.19.14.3357. PMID 11454883
- [Background] Dombernowsky P, Smith I, Falkson G, Leonard R, Panasci L, Bellmunt J, Bezwoda W, Gardin G, Gudgeon A, Morgan M, Fornasiero A, Hoffmann W, Michel J, Hatschek T, Tjabbes T, Chaudri HA, Hornberger U, Trunet PF. Letrozole, a new oral aromatase inhibitor for advanced breast cancer: double-blind randomized trial showing a dose effect and improved efficacy and tolerability compared with megestrol acetate. J Clin Oncol. 1998 Feb;16(2):453-61. doi: 10.1200/JCO.1998.16.2.453. PMID 9469328
- [Background] Bonneterre J, Buzdar A, Nabholtz JM, Robertson JF, Thurlimann B, von Euler M, Sahmoud T, Webster A, Steinberg M; Arimidex Writing Committee; Investigators Committee Members. Anastrozole is superior to tamoxifen as first-line therapy in hormone receptor positive advanced breast carcinoma. Cancer. 2001 Nov 1;92(9):2247-58. doi: 10.1002/1097-0142(20011101)92:93.0.co;2-y. PMID 11745278
- [Background] Mouridsen H, Gershanovich M, Sun Y, Perez-Carrion R, Boni C, Monnier A, Apffelstaedt J, Smith R, Sleeboom HP, Janicke F, Pluzanska A, Dank M, Becquart D, Bapsy PP, Salminen E, Snyder R, Lassus M, Verbeek JA, Staffler B, Chaudri-Ross HA, Dugan M. Superior efficacy of letrozole versus tamoxifen as first-line therapy for postmenopausal women with advanced breast cancer: results of a phase III study of the International Letrozole Breast Cancer Group. J Clin Oncol. 2001 May 15;19(10):2596-606. doi: 10.1200/JCO.2001.19.10.2596. PMID 11352951
- [Background] Howell A, Robertson JF, Quaresma Albano J, Aschermannova A, Mauriac L, Kleeberg UR, Vergote I, Erikstein B, Webster A, Morris C. Fulvestrant, formerly ICI 182,780, is as effective as anastrozole in postmenopausal women with advanced breast cancer progressing after prior endocrine treatment. J Clin Oncol. 2002 Aug 15;20(16):3396-403. doi: 10.1200/JCO.2002.10.057. PMID 12177099
- [Background] Osborne CK, Pippen J, Jones SE, Parker LM, Ellis M, Come S, Gertler SZ, May JT, Burton G, Dimery I, Webster A, Morris C, Elledge R, Buzdar A. Double-blind, randomized trial comparing the efficacy and tolerability of fulvestrant versus anastrozole in postmenopausal women with advanced breast cancer progressing on prior endocrine therapy: results of a North American trial. J Clin Oncol. 2002 Aug 15;20(16):3386-95. doi: 10.1200/JCO.2002.10.058. PMID 12177098
- [Background] Howell A, Osborne CK, Morris C, Wakeling AE. ICI 182,780 (Faslodex): development of a novel, "pure" antiestrogen. Cancer. 2000 Aug 15;89(4):817-25. doi: 10.1002/1097-0142(20000815)89:43.0.co;2-6. PMID 10951345
- [Background] Robertson JF, Nicholson RI, Bundred NJ, Anderson E, Rayter Z, Dowsett M, Fox JN, Gee JM, Webster A, Wakeling AE, Morris C, Dixon M. Comparison of the short-term biological effects of 7alpha-[9-(4,4,5,5,5-pentafluoropentylsulfinyl)-nonyl]estra-1,3,5, (10)-triene-3,17beta-diol (Faslodex) versus tamoxifen in postmenopausal women with primary breast cancer. Cancer Res. 2001 Sep 15;61(18):6739-46. PMID 11559545
- [Background] Wakeling AE, Dukes M, Bowler J. A potent specific pure antiestrogen with clinical potential. Cancer Res. 1991 Aug 1;51(15):3867-73. PMID 1855205
- [Background] Mauriac L, Pippen JE, Quaresma Albano J, Gertler SZ, Osborne CK. Fulvestrant (Faslodex) versus anastrozole for the second-line treatment of advanced breast cancer in subgroups of postmenopausal women with visceral and non-visceral metastases: combined results from two multicentre trials. Eur J Cancer. 2003 Jun;39(9):1228-33. doi: 10.1016/s0959-8049(03)00199-0. PMID 12763210
- [Background] Addo S, Yates RA, Laight A. A phase I trial to assess the pharmacology of the new oestrogen receptor antagonist fulvestrant on the endometrium in healthy postmenopausal volunteers. Br J Cancer. 2002 Dec 2;87(12):1354-9. doi: 10.1038/sj.bjc.6600644. PMID 12454761
- [Background] DeFriend DJ, Anderson E, Bell J, Wilks DP, West CM, Mansel RE, Howell A. Effects of 4-hydroxytamoxifen and a novel pure antioestrogen (ICI 182780) on the clonogenic growth of human breast cancer cells in vitro. Br J Cancer. 1994 Aug;70(2):204-11. doi: 10.1038/bjc.1994.281. PMID 8054267
- [Background] Brueggemeier RW, Hackett JC, Diaz-Cruz ES. Aromatase inhibitors in the treatment of breast cancer. Endocr Rev. 2005 May;26(3):331-45. doi: 10.1210/er.2004-0015. Epub 2005 Apr 6. PMID 15814851
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Coombes RC, Hall E, Gibson LJ, Paridaens R, Jassem J, Delozier T, Jones SE, Alvarez I, Bertelli G, Ortmann O, Coates AS, Bajetta E, Dodwell D, Coleman RE, Fallowfield LJ, Mickiewicz E, Andersen J, Lonning PE, Cocconi G, Stewart A, Stuart N, Snowdon CF, Carpentieri M, Massimini G, Bliss JM, van de Velde C; Intergroup Exemestane Study. A randomized trial of exemestane after two to three years of tamoxifen therapy in postmenopausal women with primary breast cancer. N Engl J Med. 2004 Mar 11;350(11):1081-92. doi: 10.1056/NEJMoa040331. PMID 15014181
- [Background] Howell A, Cuzick J, Baum M, Buzdar A, Dowsett M, Forbes JF, Hoctin-Boes G, Houghton J, Locker GY, Tobias JS; ATAC Trialists' Group. Results of the ATAC (Arimidex, Tamoxifen, Alone or in Combination) trial after completion of 5 years' adjuvant treatment for breast cancer. Lancet. 2005 Jan 1-7;365(9453):60-2. doi: 10.1016/S0140-6736(04)17666-6. PMID 15639680
- [Background] Kao YC, Cam LL, Laughton CA, Zhou D, Chen S. Binding characteristics of seven inhibitors of human aromatase: a site-directed mutagenesis study. Cancer Res. 1996 Aug 1;56(15):3451-60. PMID 8758911
- [Background] Johnston SR, Dowsett M. Aromatase inhibitors for breast cancer: lessons from the laboratory. Nat Rev Cancer. 2003 Nov;3(11):821-31. doi: 10.1038/nrc1211. No abstract available. PMID 14668813
- [Background] Sourdaine P, Parker MG, Telford J, Miller WR. Analysis of the aromatase cytochrome P450 gene in human breast cancers. J Mol Endocrinol. 1994 Dec;13(3):331-7. doi: 10.1677/jme.0.0130331. PMID 7893351
- [Background] Miller WR. Biological rationale for endocrine therapy in breast cancer. Best Pract Res Clin Endocrinol Metab. 2004 Mar;18(1):1-32. doi: 10.1016/s1521-690x(03)00044-7. PMID 14687595
- [Background] Jeng MH, Shupnik MA, Bender TP, Westin EH, Bandyopadhyay D, Kumar R, Masamura S, Santen RJ. Estrogen receptor expression and function in long-term estrogen-deprived human breast cancer cells. Endocrinology. 1998 Oct;139(10):4164-74. doi: 10.1210/endo.139.10.6229. PMID 9751496
- [Background] Shim WS, Conaway M, Masamura S, Yue W, Wang JP, Kmar R, Santen RJ. Estradiol hypersensitivity and mitogen-activated protein kinase expression in long-term estrogen deprived human breast cancer cells in vivo. Endocrinology. 2000 Jan;141(1):396-405. doi: 10.1210/endo.141.1.7270. PMID 10614662
- [Background] Chan CM, Martin LA, Johnston SR, Ali S, Dowsett M. Molecular changes associated with the acquisition of oestrogen hypersensitivity in MCF-7 breast cancer cells on long-term oestrogen deprivation. J Steroid Biochem Mol Biol. 2002 Aug;81(4-5):333-41. doi: 10.1016/s0960-0760(02)00074-2. PMID 12361723
- [Background] Martin LA, Farmer I, Johnston SR, Ali S, Marshall C, Dowsett M. Enhanced estrogen receptor (ER) alpha, ERBB2, and MAPK signal transduction pathways operate during the adaptation of MCF-7 cells to long term estrogen deprivation. J Biol Chem. 2003 Aug 15;278(33):30458-68. doi: 10.1074/jbc.M305226200. Epub 2003 May 29. PMID 12775708
- [Background] Santen RJ, Song RX, Zhang Z, Kumar R, Jeng MH, Masamura S, Lawrence J Jr, MacMahon LP, Yue W, Berstein L. Adaptive hypersensitivity to estrogen: mechanisms and clinical relevance to aromatase inhibitor therapy in breast cancer treatment. J Steroid Biochem Mol Biol. 2005 May;95(1-5):155-65. doi: 10.1016/j.jsbmb.2005.04.025. PMID 16024245
- [Background] Borras M, Laios I, el Khissiin A, Seo HS, Lempereur F, Legros N, Leclercq G. Estrogenic and antiestrogenic regulation of the half-life of covalently labeled estrogen receptor in MCF-7 breast cancer cells. J Steroid Biochem Mol Biol. 1996 Feb;57(3-4):203-13. doi: 10.1016/0960-0760(95)00272-3. PMID 8645630
- [Background] Dauvois S, White R, Parker MG. The antiestrogen ICI 182780 disrupts estrogen receptor nucleocytoplasmic shuttling. J Cell Sci. 1993 Dec;106 ( Pt 4):1377-88. doi: 10.1242/jcs.106.4.1377. PMID 8126115
- [Background] Ingle JN, Suman VJ, Rowland KM, Mirchandani D, Bernath AM, Camoriano JK, Fishkin PA, Nikcevich DA, Perez EA; North Central Cancer Treatment Group Trial N0032. Fulvestrant in women with advanced breast cancer after progression on prior aromatase inhibitor therapy: North Central Cancer Treatment Group Trial N0032. J Clin Oncol. 2006 Mar 1;24(7):1052-6. doi: 10.1200/JCO.2005.04.1053. PMID 16505423
- [Background] Perey L, Paridaens R, Hawle H, Zaman K, Nole F, Wildiers H, Fiche M, Dietrich D, Clement P, Koberle D, Goldhirsch A, Thurlimann B. Clinical benefit of fulvestrant in postmenopausal women with advanced breast cancer and primary or acquired resistance to aromatase inhibitors: final results of phase II Swiss Group for Clinical Cancer Research Trial (SAKK 21/00). Ann Oncol. 2007 Jan;18(1):64-69. doi: 10.1093/annonc/mdl341. Epub 2006 Oct 9. PMID 17030543
- [Background] Gradishar WJ, Sahmoud T. Current and future perspectives on fulvestrant. Clin Breast Cancer. 2005 Apr;6 Suppl 1:S23-9. doi: 10.3816/cbc.2005.s.011. PMID 15865847
- [Background] McClelland RA, Barrow D, Madden TA, Dutkowski CM, Pamment J, Knowlden JM, Gee JM, Nicholson RI. Enhanced epidermal growth factor receptor signaling in MCF7 breast cancer cells after long-term culture in the presence of the pure antiestrogen ICI 182,780 (Faslodex). Endocrinology. 2001 Jul;142(7):2776-88. doi: 10.1210/endo.142.7.8259. PMID 11415996
- [Background] Cockerill S, Stubberfield C, Stables J, Carter M, Guntrip S, Smith K, McKeown S, Shaw R, Topley P, Thomsen L, Affleck K, Jowett A, Hayes D, Willson M, Woollard P, Spalding D. Indazolylamino quinazolines and pyridopyrimidines as inhibitors of the EGFr and C-erbB-2. Bioorg Med Chem Lett. 2001 Jun 4;11(11):1401-5. doi: 10.1016/s0960-894x(01)00219-0. PMID 11378364
- [Background] Xia W, Mullin RJ, Keith BR, Liu LH, Ma H, Rusnak DW, Owens G, Alligood KJ, Spector NL. Anti-tumor activity of GW572016: a dual tyrosine kinase inhibitor blocks EGF activation of EGFR/erbB2 and downstream Erk1/2 and AKT pathways. Oncogene. 2002 Sep 12;21(41):6255-63. doi: 10.1038/sj.onc.1205794. PMID 12214266
- [Background] Rusnak DW, Lackey K, Affleck K, Wood ER, Alligood KJ, Rhodes N, Keith BR, Murray DM, Knight WB, Mullin RJ, Gilmer TM. The effects of the novel, reversible epidermal growth factor receptor/ErbB-2 tyrosine kinase inhibitor, GW2016, on the growth of human normal and tumor-derived cell lines in vitro and in vivo. Mol Cancer Ther. 2001 Dec;1(2):85-94. PMID 12467226
- [Background] Holbro T, Beerli RR, Maurer F, Koziczak M, Barbas CF 3rd, Hynes NE. The ErbB2/ErbB3 heterodimer functions as an oncogenic unit: ErbB2 requires ErbB3 to drive breast tumor cell proliferation. Proc Natl Acad Sci U S A. 2003 Jul 22;100(15):8933-8. doi: 10.1073/pnas.1537685100. Epub 2003 Jul 9. PMID 12853564